CLINICAL TRIAL: NCT00069719
Title: Phase II Safety and Efficacy Study to Evaluate a Glaucoma Therapy in Open-Angle Glaucoma or Ocular Hypertension Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-33; C-02-33
Record Dates: First submitted 2003-09-30; First posted 2003-10-06 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: open-angle; glaucoma; ocular; hypertension; POAG
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension

INTERVENTIONS:
Drug: Glaucoma therapy

SUMMARY:
To determine the safety and IOP-lowering ability of a test compound in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects of either sex and any race with open-angle glaucoma or ocular hypertension;
* logMAR visual acuity not worse than 0.6.

Exclusion Criteria:

* Clinically relevant ophthalmic or systemic conditions may be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Clinical Trial Sites, Multiple Locations Throughout the US Sponsored by Alcon of, Texas, United States